CLINICAL TRIAL: NCT05877573
Title: Toripalimab Combined With Neoadjuvant Chemoradiotherapy as First-line Treatment for Locally Advanced，High-Risk，MSS Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-062
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced; High-Risk; Rectal Cancer; MSS
MeSH Terms: conditions — Rectal Neoplasms | interventions — toripalimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- short-course radiotherapy plus chemotherapy and immunotherapy (Experimental): A total of 53 patients receive 5*5Gy short-course radiotherapy, followed by 4 cycles of CAPOX chemotherapy and PD-1 antibody, finally receive the TME surgery and another 2 cycles of CAPOX chemotherapy.
  Interventions: Drug: Toripalimab; Radiation: short-term radiotherapy; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg,d1,q3w
Radiation: short-term radiotherapy — 25Gy/5Fx
  Other Names: shor-course radiotherapy
Drug: Oxaliplatin — 135mg/m2 d1 q3w
Drug: Capecitabine — 1200mg/m2 d1-14 q3w

SUMMARY:
This is a single arm, open-label, prospective clinical trial to evaluate the combination of neoadjuvant short-course radiotherapy and toripalimab (PD-1 antibody) for locally advanced rectal cancer (LARC) patients with high risk factors. A total of 53patients will be enrolled in this trial to receive 5*5Gy short-course radiotherapy, followed by 4 cycles of CAPOX chemotherapy and PD-1 antibody. Then they will receive the TME surgery and another 2 cycles of CAPOX chemotherapy. The primary end point is the rate of pathological complete response (pCR). The long-term prognosis and adverse effects will also be evaluated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, female and male;
* Pathological confirmed MSS or pMMR rectal adenocarcinoma;
* Clinical stage T3-4 (AJCC 8th) and at least with one high risk factor（CRM+ or EMVI+ or lateral lymph nodes+）;
* No previous chemotherapy, radiotherapy, immunotherapy or other anti-tumor treatment;
* Adequate organ function defined at baseline as:

ANC ≥1.5××109/L，PLt ≥100×109 /L，Hb ≥90 g/L，15×109 /L≥WBC≥4×109 /L; TBIL ≤1.5×ULN, ALT ≤1.5ULN, AST ≤1.5ULN, BUN and Cr ≤1.5×ULN or Ccr

* 60ml/min (Cockcroft-Gault formula);INR ≤1.5×ULN or PT ≤1.5×ULN (when patient didn't accept anticoagulant therapy);

  * Women of childbearing age must have taken reliable contraceptive measures or have a pregnancy test (serum or urine) within 7 days prior to enrollment and the results are negative;

Exclusion Criteria:

* Pathological confirmed rectal squamous cell carcinoma;
* History of other uncured malignancies within 5 years;
* Allergic to any component of chemotherapy or immunotherapy;
* History of any active, known, or suspected autoimmune disease, including but not limited to myasthenia gravis,Myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis,Inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulation Swollen disease, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis or Glomerulonephritis.
* With congenital or acquired immunodeficiency (such as those with HIV infection), active hepatitis B or hepatitis C;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | The TME surgery will be recommended after the neoadjuvant therapy. The pCR rate is evaluated after surgery. Assessed up to 6 months
  Pathologic complete response rate

SECONDARY OUTCOMES:
3-year ORR | Assessed up to 3 years
  3-year objective response rate
3-year DCR | Assessed up to 3 years
  3-year disease control rate
3-year OS | Assessed up to 3 years
  3-year overall survival rate
AE | Assessed up to 3 years
  adverse event
SAE | Assessed up to 3 years
  Serious Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Dehua Wu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No